CLINICAL TRIAL: NCT04089072
Title: Methylene Blue as a Third-line Vasopressor in Septic Shock to Maintain Hemodynamics
Brief Title: Methylene Blue as a Third-line Vasopressor in Septic Shock
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carilion Clinic (Other)
Collaborators: Provepharm Life Solutions (Unknown)
Responsible Party: Principal Investigator, Frank H Biscardi, MD, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 19-549
Record Dates: First submitted 2019-08-23; First posted 2019-09-13 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Septic Shock
Keywords: Methylene Blue; Vasopressors; Septic Shock; Provay Blue®
MeSH Terms: conditions — Shock, Septic | interventions — Methylene Blue; Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Experimental): Patients in the control group will have phenylephrine infusion starting at 50 mcg/min and titrated to maintain a MAP >65 mmHg as a third line vasopressor. Maximum dose of Phenylephrine is 300 mcg/min.
  Interventions: Drug: Phenylephrine
- Intervention group (Experimental): Patients enrolled in the intervention group will receive 2 mg/kg IBW (Ideal Body Weight) bolus, given over 15 mins, of ProvayBlue® followed by a concomitant infusion at 2 mg/kg/hr (IBW) mixed in D5W, which will continue for 24 hours. ProvayBlue® ( Methylene Blue) will be used as the third-line vasopressor.
  Interventions: Drug: Methylene Blue

INTERVENTIONS:
Drug: Methylene Blue — Prior to the initiation of the randomized treatment, the subject will have received 2 vasopressors ( norepinephrine and vasopressin), they will be initiated on IV hydrocortisone . Once the patient is unable to maintain a mean arterial pressure of >65mmHg and the hydrocortisone has been administered there will be an addition of a third-line vasopressor.
  Patients enrolled in the intervention group will receive ProvayBlue® and Patients enrolled in the control group will receive Phenylephrine infusion as a third line vasopressor in the treatment of septic shock.
  Other Names: ProvayBlue®
  Arms: Intervention group
Drug: Phenylephrine — Prior to the initiation of the randomized treatment, the subject will have received 2 vasopressors ( norepinephrine and vasopressin) already , they will be initiated on IV hydrocortisone . Once the patient is unable to maintain a mean arterial pressure of >65mmHg and the hydrocortisone has been administered there will be an addition of a third-line vasopressor.
  Patients enrolled in the intervention group will receive ProvayBlue® and Patients enrolled in the control group will receive Phenylephrine infusion as a third line vasopressor in the treatment of septic shock.
  Arms: Control group

SUMMARY:
A randomized, prospective study comparing ProvayBlue® to standard care with multiple sympathomimetic vasopressors.

DETAILED DESCRIPTION:
The study will be an un-blinded, Phase 2, randomized, 1:1, prospective trial comparing patients in septic shock receiving norepinephrine and vasopressin followed by phenylephrine versus ProvayBlue® as the third-line vasopressor. The third line vasopressor will be compared at 1 hour to see if it affects the patient's mean arterial blood pressure (MAP).

ELIGIBILITY:
Inclusion Criteria:

1. Meets Sepsis-3 Criteria (Suspected source of infection plus any 2 criteria of the qSOFA)

2 .Septic Shock (any patient requiring vasopressor therapy to maintain MAP >65 mmHg or any patient with serum lactate >2 mmol/dL even in the absence of hypovolemia ).

3) Greater than 18 years old

4 ) ICU Admission

Exclusion Criteria:

Inability to obtain informed consent from an appropriate surrogate decision maker.

Also:

1. Children less than 18 years old
2. Pregnant women or positive urinary pregnancy test in reproductive-aged women
3. Prisoners
4. Evolving myocardial infarction or known cardiomyopathy with documented EF<35%
5. Known grade 3 diastolic dysfunction document by echocardiogram
6. Known hypersensitivity to thiazine dyes
7. Pulmonary hypertension that is currently requiring vasodilator therapy
8. Concurrent form of shock present or suspected: Obstructive, Neurogenic, Hemorrhagic
9. Known documented history of G6PD deficiency or favism
10. Active prior to admission medication prescription for a SSRI or SNRI , systemic heparin anticoagulation or other medications listed above (under Study Agent). These medications will be listed in the printed enrollment form.
11. Severe renal failure is a contraindication to use of ProvayBlue®.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in mean arterial pressure | One hour and 24 hours after dose
  The primary objective is to determine if the administration of ProvayBlue® is non-inferior to the use of phenylephrine as a third-line vasopressor to keep a mean arterial pressure (MAP)>65 mmhg after one hour and at 24 hours after the initiation of the drugs.

SECONDARY OUTCOMES:
Incidence of acute kidney injury requiring dialysis | through time of patient discharge, an average of 8 days after admission
  The secondary objectives are to see if the total vasopressor dosing and renal replacement needs are different in those patients receiving ProvayBlue® rather than standard care with escalating number of vasopressors.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Biscardi, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
To publish aggregated data